CLINICAL TRIAL: NCT07147491
Title: Study to Verify the Effectiveness and Safety of the Electrically Powered Orthopedic Exercise Device on Gait Ability in Patients Who Have Undergone Hip Surgery: Investigator-Initiated, Single-Center, Single-Group Clinical Trial
Brief Title: Effectiveness and Safety of the Electrically Powered Orthopedic Exercise Device on Gait Ability in Patients With Who Have Undergone Hip Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9-2025-0017
Record Dates: First submitted 2025-04-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hip Surgery
Keywords: Rehabilitation; Gait; Wearable robot; Hip Surgery

STUDY DESIGN:
Intervention Model Description: Researchers will compare non-wearing and wearing conditions of the electrically powered orthopedic exercise device walking speeds, spatiotemporal parameters, balance in participants and does not establish a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearing conditions of Electrically Powered Orthopedic Exercise Device (Experimental): Participants will undergo gait and balance function tests under both non-wearing and wearing conditions of the electrically powered orthopedic exercise device
  Interventions: Device: Electrically Powered Orthopedic Exercise Device

INTERVENTIONS:
Device: Electrically Powered Orthopedic Exercise Device — Participants who pass the screening undergo an evaluation of gait function and balance ability without wearing the Electrically Powered Orthopedic Exercise Device. Afterward, the patient wears the motorized orthopedic exercise device for a total of four adaptation sessions. In each session, the patient performs short-distance walking within 10 meters while wearing the device to explore the appropriate assistive mode and level of support that match their physical condition. No evaluations are conducted while wearing the device during sessions 1, 2, and 3. After the 4th session, an evaluation identical to the one conducted without the device is performed while wearing it, and a satisfaction survey is conducted.

SUMMARY:
Gait is an essential daily activity performed through the complex coordination of the central and peripheral nervous systems and the musculoskeletal system. Gait disorders can negatively affect quality of life, increase the risk of falls, decrease the ability to perform daily activities, and limit physical activity. Gait disorders can result from various musculoskeletal conditions, with hip osteoarthritis, avascular necrosis of the femoral head, and hip fractures being the most representative causes.

In the early stages of hip osteoarthritis, avascular necrosis of the femoral head, or non-severely displaced hip fractures, various intervention therapies, including rehabilitation exercise therapy and injection treatments, can be attempted. However, these intervention therapies only alleviate symptoms and cannot prevent disease progression. Consequently, most patients eventually experience thinning of the full-thickness hip cartilage, collapse of the femoral head, nonunion, or worsening displacement, which leads to restricted hip range of motion. As a result, lower limb muscle weakness and functional decline occur, ultimately requiring hip surgeries such as total hip arthroplasty or open reduction and internal fixation. Although most patients experience a recovery in gait ability after hip surgery, some show a slower recovery rate or fail to achieve normal walking.

It has been reported that over 80% of function is recovered by three months after surgery; however, during this period, patients experience limitations in performing daily activities. As a compensatory mechanism, excessive weight-bearing on the non-operated limb may occur, increasing the risk of overloading the non-operated hip. This may lead to the development of osteoarthritis in the non-operated limb and has also been reported to increase the risk of falls. Therefore, various methods are being studied to facilitate gait function recovery after hip surgery and promote an early return to daily activities.

Therefore, this study aims to explore the clinical feasibility of the Angel Suit H10 (Angelrobotics, Seoul, Korea) by assessing whether wearing the Electrically Powered Orthopedic Exercise Device improves gait function in patients who have undergone hip surgery, along with evaluating user satisfaction and device safety.

DETAILED DESCRIPTION:
(1) Overview of study design This investigator-initiated exploratory study is a pilot study designed to evaluate the effectiveness and safety of the Electrically Powered Orthopedic Exercise Device by measuring and analyzing gait function and balance ability in patients who have undergone hip surgery under both non-wearing and wearing conditions.

(2) Experimental Group and Evaluation Procedures

1. Participant Selection:

   This study includes a single test group with a total of 30 participants. The selection of participants for the electrically powered orthopedic exercise device and the overall study process will be conducted under the prescription and guidance of a rehabilitation medicine specialist, and supervised by assistants (physicians and occupational therapists). The examiner will collect clinical information and conduct a screening assessment for each participant.
2. Evaluation Phase Without Device:

   After the screening test, participants undergo assessments of walking ability and balance without wearing the motorized orthopedic exercise device. A 10-minute rest period is provided between each assessment. If the participant wishes, additional rest time is allowed and recorded in the case report form. The assessments include the 10-Meter Walk Test, the 6-Minute Walk Test, the Timed Up and Go Test, and the Berg Balance Scale. These evaluations are conducted in the rehabilitation function testing room on the second floor of the facility under the supervision of the research team (physician and either a physical or occupational therapist).
3. Pre-Adaptation Phase:

   After the evaluations without the device, a total of four adaptation sessions are conducted, during which the participant wears the device and performs short-distance walking within 10 meters. These sessions are designed to help the participant become familiar with the operation and wearing method of the H10 device. Appropriate device settings are configured for each participant to minimize any potential inexperience or anxiety during use. Participants must complete all four adaptation sessions, and each session should be conducted within a two-week interval.
4. Evaluation Phase:

After completing all four adaptation sessions, participants undergo assessments of walking ability and balance while wearing the motorized orthopedic exercise device. A 10-minute rest period is provided between each assessment. If the participant wishes, additional rest time is allowed and recorded in the case report form. The assessments include the 10-Meter Walk Test, the 6-Minute Walk Test, the Timed Up and Go Test, and the Berg Balance Scale. These evaluations are conducted in the rehabilitation function testing room on the second floor of the facility under the supervision of the research team (physician and either a physical or occupational therapist). After the evaluations are completed, a usability and satisfaction survey regarding the motorized orthopedic exercise device is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 19 or older
2. Individuals who have undergone hip surgery due to hip osteoarthritis, avascular necrosis of the femoral head, or hip fracture
3. Individuals who are at least two days post-hip surgery and are assessed to be medically stable
4. Individuals who have adequate cognitive ability (Korean Mini-Mental State Examination score ≥ 20)
5. Individuals able to sit at the edge of a bed without assistance and stand for 10 seconds regardless of support
6. Individuals who are Functional Ambulatory Category (FAC) score of 1-3
7. Individuals who visited Yongin Severance Hospital, understood the study, and signed informed consent

Exclusion Criteria:

1. Individuals who, after undergoing hip surgery, present with exudate at the surgical site or report symptoms such as heat, redness, swelling, or severe pain at the affected area
2. Individuals who have contraindications for lower limb weight-bearing such as severe joint contractures, osteoporosis, or untreated fractures
3. Individuals who have progressive or unstable brain diseases or neurological paralysis from stroke
4. Individuals who have active infections or open wounds hindering device use
5. Individuals who have significant leg length discrepancies
6. Individuals who have severe deformities or contractures in the lower extremities
7. Individuals who have history of poliomyelitis
8. Individuals inable to maintain seated or standing positions independently
9. Individuals who have severe spasticity (Modified Ashworth Scale grade ≥ 2)
10. Individuals who have bone metastases from cancer
11. Individuals who have severe internal diseases affecting device use (e.g., cardiovascular or respiratory diseases)
12. Individuals who have cognitive impairments preventing cooperation with device use
13. Individuals who have complaints of device-related side effects or potential rehabilitation discontinuation (e.g., severe obesity, skeletal deformity)
14. Patients who are determined to be pregnant or potentially pregnant based on the medical interview
15. Individuals who have any other clinically significant findings deemed inappropriate by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
10-Meter Walk Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are instructed to walk 14 m, including 2 m at both ends for acceleration and deceleration, at their comfortable speed. Gait speed was calculated by dividing the 10m distance by the time taken.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Researchers ask patients to rise from a seated position, walk a distance of 3 m, turn around, return to the chair, and sit back. The average time of three trials was recorded as a result
6-Minute Walk Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are instructed to walk back and forth along the 30-meter path as many times as possible within 6 minutes. The examiner records the total distance covered, abnormal gait patterns, and the time of occurrence of any gait deviations.
Berg balance scale (BBS) | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are asked to perform 14 tasks regarding the static and dynamic balance of patients. Each task was rated on a five-point scale from 0 to 4, with a total score of 56.
Spatiotemporal Parameters of Gait : Total Step Count | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Total Step Count: The total number of steps taken during walking.
Spatiotemporal Parameters of Gait : Cadence | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Cadence: The number of steps taken per minute, measured in steps per minute (spm).
Spatiotemporal Parameters of Gait : Self-Selected Walking Speed | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Self-Selected Walking Speed: The participant's walking speed when walking naturally at a comfortable pace.
Spatiotemporal Parameters of Gait : Distance | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Distance: The total distance covered during walking, measured in meters (m).
Spatiotemporal Parameters of Gait : Stride Length | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Stride Length: The distance between the heel of one foot to the heel of the same foot during consecutive steps. Measured in meters (m), stride length is adjusted for height to account for differences in body size.
Satisfaction evaluation | Upon completion of the end-point assessment conducted on the same day as session 4
  Participants will complete a satisfaction survey for usability and satisfaction assessment of the electrically powered orthopedic exercise device, based on the Korean version of the Quebec User Evaluation of Satisfaction with assistive Technology (K-QUEST 2.0).21 This survey consists of 12 items on a 5-point scale. Participants rate their satisfaction with the assistive device and related services

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee, Sang-Heon, Bong-Keun Jung, and So-Yeon Park. "Korean Translation and Psychometric Properties of Quebec User Evaluation of Satisfaction Assistive Technology 2.0." Journal of the Korea Academia-Industrial Cooperation Society. The Korea Academia-Industrial Cooperation Society, July 31, 2013.
- [Background] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Background] Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Berman LB. The 6-minute walk: a new measure of exercise capacity in patients with chronic heart failure. Can Med Assoc J. 1985 Apr 15;132(8):919-23. PMID 3978515
- [Background] Hwang R, Morris NR, Mandrusiak A, Mudge A, Suna J, Adsett J, Russell T. Timed Up and Go Test: A Reliable and Valid Test in Patients With Chronic Heart Failure. J Card Fail. 2016 Aug;22(8):646-50. doi: 10.1016/j.cardfail.2015.09.018. Epub 2015 Oct 9. PMID 26456063
- [Background] Santos M, Zdravevski E, Albuquerque C, Coelho PJ, Pires IM. Ten Meter Walk Test for motor function assessment with technological devices based on lower members' movements: A systematic review. Comput Biol Med. 2025 Mar;187:109734. doi: 10.1016/j.compbiomed.2025.109734. Epub 2025 Feb 3. PMID 39904103
- [Background] Kim Heon-tae, Moon Jun-bae, Ryu Seung-ho, and Kang Min-soo. Validity study of the Korean version of the International Physical Activity Questionnaire (IPAQ): Verification of construct-related validity. Korean Journal of Physical Education No. 2017;56
- [Background] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114
- [Background] Cuthbert SC, Goodheart GJ Jr. On the reliability and validity of manual muscle testing: a literature review. Chiropr Osteopat. 2007 Mar 6;15:4. doi: 10.1186/1746-1340-15-4. PMID 17341308
- [Background] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Background] Kang Y, NA D-L, Hahn S. A validity study on the Korean Mini-Mental State Examination (K-MMSE) in dementia patients. Journal of the Korean neurological association 1997:300-308
- [Background] Ikutomo H, Nagai K, Nakagawa N, Masuhara K. Falls in patients after total hip arthroplasty in Japan. J Orthop Sci. 2015 Jul;20(4):663-8. doi: 10.1007/s00776-015-0715-7. Epub 2015 Mar 24. PMID 25797333
- [Background] Smith TO, Pearson M, Latham SK. Are people following hip and knee arthroplasty at greater risk of experiencing a fall and fracture? Data from the Osteoarthritis Initiative. Arch Orthop Trauma Surg. 2016 Jun;136(6):865-72. doi: 10.1007/s00402-016-2445-5. Epub 2016 Mar 19. PMID 26994762
- [Background] Suter E, Herzog W, Leonard TR, Nguyen H. One-year changes in hind limb kinematics, ground reaction forces and knee stability in an experimental model of osteoarthritis. J Biomech. 1998 Jun;31(6):511-7. doi: 10.1016/s0021-9290(98)00041-4. PMID 9755035
- [Background] Abujaber S, Pozzi F, Zeni J Jr. Influence of weight bearing visual feedback on movement symmetry during sit to stand task. Clin Biomech (Bristol). 2017 Aug;47:110-116. doi: 10.1016/j.clinbiomech.2017.06.005. Epub 2017 Jun 8. PMID 28641199
- [Background] Abujaber SB, Marmon AR, Pozzi F, Rubano JJ, Zeni JA Jr. Sit-To-Stand Biomechanics Before and After Total Hip Arthroplasty. J Arthroplasty. 2015 Nov;30(11):2027-33. doi: 10.1016/j.arth.2015.05.024. Epub 2015 May 19. PMID 26117068
- [Background] Miura N, Tagomori K, Ikutomo H, Nakagawa N, Masuhara K. Asymmetrical loading during sit-to-stand movement in patients 1 year after total hip arthroplasty. Clin Biomech (Bristol). 2018 Aug;57:89-92. doi: 10.1016/j.clinbiomech.2018.06.017. Epub 2018 Jun 25. PMID 29966959
- [Background] McCrory JL, White SC, Lifeso RM. Vertical ground reaction forces: objective measures of gait following hip arthroplasty. Gait Posture. 2001 Oct;14(2):104-9. doi: 10.1016/s0966-6362(01)00140-0. PMID 11544061
- [Background] Talis VL, Grishin AA, Solopova IA, Oskanyan TL, Belenky VE, Ivanenko YP. Asymmetric leg loading during sit-to-stand, walking and quiet standing in patients after unilateral total hip replacement surgery. Clin Biomech (Bristol). 2008 May;23(4):424-33. doi: 10.1016/j.clinbiomech.2007.11.010. Epub 2007 Dec 31. PMID 18164792
- [Background] Murray MP, Brewer BJ, Zuege RC. Kinesiologic measurements of functional performance before and after McKee-Farrar total hip replacement. A study of thirty patients with rheumatoid arthritis, osteoarthritis, or avascular necrosis of the femoral head. J Bone Joint Surg Am. 1972 Mar;54(2):237-56. No abstract available. PMID 4651259
- [Background] Bennett D, Humphreys L, O'Brien S, Kelly C, Orr JF, Beverland DE. Gait kinematics of age-stratified hip replacement patients--a large scale, long-term follow-up study. Gait Posture. 2008 Aug;28(2):194-200. doi: 10.1016/j.gaitpost.2007.11.010. Epub 2008 Feb 19. PMID 18242996
- [Background] Organisation for Economic Co-operation and Development. OECD Health Data. 2017. http://dx.doi.org/10.1787/888933605236
- [Background] Kinds MB, Welsing PM, Vignon EP, Bijlsma JW, Viergever MA, Marijnissen AC, Lafeber FP. A systematic review of the association between radiographic and clinical osteoarthritis of hip and knee. Osteoarthritis Cartilage. 2011 Jul;19(7):768-78. doi: 10.1016/j.joca.2011.01.015. Epub 2011 Jan 31. PMID 21281726
- [Background] Murphy NJ, Eyles JP, Hunter DJ. Hip Osteoarthritis: Etiopathogenesis and Implications for Management. Adv Ther. 2016 Nov;33(11):1921-1946. doi: 10.1007/s12325-016-0409-3. Epub 2016 Sep 26. PMID 27671326
- [Background] Alves EM, Angrisani AT, Santiago MB. The use of extracorporeal shock waves in the treatment of osteonecrosis of the femoral head: a systematic review. Clin Rheumatol. 2009 Nov;28(11):1247-51. doi: 10.1007/s10067-009-1231-y. Epub 2009 Jul 17. PMID 19609482
- [Background] Bennell KL, Buchbinder R, Hinman RS. Physical therapies in the management of osteoarthritis: current state of the evidence. Curr Opin Rheumatol. 2015 May;27(3):304-11. doi: 10.1097/BOR.0000000000000160. PMID 25775185
- [Background] Gay C, Chabaud A, Guilley E, Coudeyre E. Educating patients about the benefits of physical activity and exercise for their hip and knee osteoarthritis. Systematic literature review. Ann Phys Rehabil Med. 2016 Jun;59(3):174-183. doi: 10.1016/j.rehab.2016.02.005. Epub 2016 Apr 1. PMID 27053003
- [Background] Paans N, van den Akker-Scheek I, Dilling RG, Bos M, van der Meer K, Bulstra SK, Stevens M. Effect of exercise and weight loss in people who have hip osteoarthritis and are overweight or obese: a prospective cohort study. Phys Ther. 2013 Feb;93(2):137-46. doi: 10.2522/ptj.20110418. Epub 2012 Sep 27. PMID 23023813
- [Background] Alexander NB. Gait disorders in older adults. J Am Geriatr Soc. 1996 Apr;44(4):434-51. doi: 10.1111/j.1532-5415.1996.tb06417.x. No abstract available. PMID 8636592
- [Background] Mirelman A, Shema S, Maidan I, Hausdorff JM. Gait. Handb Clin Neurol. 2018;159:119-134. doi: 10.1016/B978-0-444-63916-5.00007-0. PMID 30482309
- [Background] Baker JM. Gait Disorders. Am J Med. 2018 Jun;131(6):602-607. doi: 10.1016/j.amjmed.2017.11.051. Epub 2017 Dec 27. PMID 29288631

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT07147491/Prot_SAP_000.pdf